CLINICAL TRIAL: NCT01599611
Title: Follow-up of Extreme Neonatal Hyperbilirubinemia in 5-10 Year Old Children: a Danish Population Based Study
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: pkv
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Neonatal Hyperbilirubinemia
Keywords: Neonatal hyperbilirubinemia; Follow-up; Motor development; Hearing; Executive function
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Exposed group: Children age 5-10 years old who had a total serum bilirubin > 450 umol/L in the neonatal period
  Interventions: Procedure: Movement assessment battery for children - 2
- Non-exposed group: Matched 1:1 to the exposed group on gender, age, gestational age and municipality of residence
  Interventions: Procedure: Movement assessment battery for children - 2

INTERVENTIONS:
Procedure: Movement assessment battery for children - 2 — A standardised test developed to identify developmental difficulties in children.
  Other Names: MABC-2

SUMMARY:
The objective of this study was to investigate whether infants with total serum bilirubin > 450 umol/L in the neonatal period and no symptoms or no more than early acute bilirubin encephalopathy develop long term sequelae with impairment of motor development, hearing and executive function compared with a control group.

DETAILED DESCRIPTION:
Children in both the exposed and the non-exposed group were examined by use of the MABC-2 and pure tone audiometry by the responsible examiner for the study, Pernille Vandborg, MD. The aim was to see whether the exposed group suffered any long term sequelae to the extreme neonatal hyperbilirubinemia, i.e. impaired motor development or hearing impairment, compared to a control group. The examinations took place at the local hospital.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age > 35 weeks
* Total serum bilirubin > 450 umol/L in the neonatal period
* Born in the period 01.01.2000 - 31.12.2005

Exclusion Criteria:

* Acute intermediate or advanced bilirubin encephalopathy

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children born in Denmark in the period 01.01.2000 - 31.12.2005 with a gestational age >= 35 weeks and a total serum bilirubin > 450 umol/L and a matched control group of children
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2010-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Motor development | Age 5-10 years
  Delayed motor development for children in the exposed group compared to children in the non-exposed group

CONTACTS AND LOCATIONS:
Overall Officials: Pernille Vandborg, MD, PhD, Principal Investigator — Børneafdelingen, Aalborg Sygehus, Denmark

REFERENCES:
- [Derived] Vandborg PK, Hansen BM, Greisen G, Mathiasen R, Kasper F, Ebbesen F. Follow-up of extreme neonatal hyperbilirubinaemia in 5- to 10-year-old children: a Danish population-based study. Dev Med Child Neurol. 2015 Apr;57(4):378-84. doi: 10.1111/dmcn.12603. Epub 2014 Oct 29. PMID 25353277
- See also: A description of the study in Danish — http://www.aalborgsygehus.rn.dk/Afdelinger/Afsnit1213/Efter+undersøgelser